CLINICAL TRIAL: NCT01056263
Title: Retrospective Observational Study Of Subjects With Cytokine-Refractory Metastatic Renal Cancer Treated With Axitinib (AG-013736) To Estimate 5-Yr Survival
Brief Title: Retrospective Observational Study To Update 5-Year Survival Of Subjects Who Participated In Axitinib Trial A4061012
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4061065
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Results first posted 2012-03-28 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Carcinoma, Renal Cell
Keywords: retrospective trial; 5-year survival; metastatic renal cancer cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-Interventional Study: Subjects participating in this observational study originally participated in study A4061012 [NCT00076011], and may have also have participated in study A4061008 [NCT00828919].
  Interventions: Drug: axitinib: observational study

INTERVENTIONS:
Drug: axitinib: observational study — Non-interventional observational study
  Other Names: AG-013736

SUMMARY:
The primary objective of this observational study is to retrospectively collect current survival data for patients originally included in axitinib A4061012 [NCT00076011] study to estimate the 5-year survival rate in subjects with metastatic renal cancer cell treated with axitinib.

DETAILED DESCRIPTION:
Subjects participating in this observational study originally participated in study A4061012 [NCT00076011], and may have also have participated in study A4061008 [NCT00828919]. Subjects participating in this observational study originally participated in study A4061012 [NCT00076011], and may have also have participated in study A4061008 [NCT00828919].

5-year survival information to be updated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects participating in this observational study originally participated in study A4061012 [NCT00076011] and may have also participated in study A4061008 [NCT00828919]

Exclusion Criteria:

* Subjects who withdrew from the original study A4061012 [NCT00076011] or the continuing access study A4061008 [NCT00828919]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects participating in this observational study originally participated in study A4061012 [NCT00076011], and may have also have participated in study A4061008 [NCT00828919].
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (5):
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Madison, Wisconsin
- Pfizer Investigational Site, Paris, France
- Pfizer Investigational Site, Hanover, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061065&StudyName=Retrospective%20Observational%20Study%20To%20Update%205-Year%20Survival%20Of%20Subjects%20Who%20Participated%20In%20Axitinib%20Trial%20A4061012

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib: The study is aimed to retrospectively update the overall survival data (5-year) collected from participants who participated to a previous completed axitinib (AG-013736) study (A4061012; NCT00076011). Part of these participants continued axitinib (AG-013736) treatment after study A4061012 closure, under the roll over study (A4061008; NCT00828919).
Period: Overall Study
Arm/Group | Axitinib
Started | 52
Completed | 0
Not Completed | 52
Not completed — Adverse Event | 12
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 29
Not completed — Progressive disease | 2
Not completed — Neoplasm progression | 1
Not completed — Objective progression or relapse | 1
Not completed — Ongoing in study A4061008 (NCT00828919) | 5

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib
Number analyzed (Participants) | 52
Age Continuous [Mean (Standard Deviation); unit: years] | 58.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is the duration from first dose of study medication to death. For participants who are alive, overall survival is censored at the last contact.
Time Frame: Baseline until death or up to Year 5
Population: Full analysis set included all participants who received at least 1 dose of axitinib (AG-013736).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 52
Days | 911.0 [670.0 to 1283.0]
Statistical Analysis 1: Comparison: Axitinib; Five year survival probability was the probability of survival at 5 year after the date of the start of the study treatment based on the Kaplan-Meier estimate; Test type: Superiority or Other; Five year survival probability = 20.60, 95% CI 2-sided [10.94 to 32.38]

ADVERSE EVENTS:
Description: There were no adverse events collected in this retrospective study.
Arm/Group | Axitinib
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.